CLINICAL TRIAL: NCT07327346
Title: Test-Retest and Interrater Reliability and Validity of Postural Sway Parameters Measured With GYKO During the L Test in Individuals With Parkinson's Disease
Brief Title: GYKO-Based L-Test Reliability in Parkinson's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Büşra Akıncı, MSc, Hasan Kalyoncu University
Other Study IDs: HKU/PH/2
Record Dates: First submitted 2025-12-08; First posted 2026-01-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; balance; postural sway; interrater reliability; test-retest reliabilit; validity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease group: Parkinson's disease patients with stage 1-3 hoehn yahr
  Interventions: Other: GYKO-Based Postural Sway Assessment

INTERVENTIONS:
Other: GYKO-Based Postural Sway Assessment — This procedure involves obtaining postural sway parameters using the GYKO inertial measurement device during the Time Up and Go (TUG) test and L-Test. No therapeutic intervention is applied.
  Time Up and Go Test: Timed Up and Go (TUG) is a standardized functional mobility test used to assess dynamic balance and gait performance. Participants are instructed to stand up from a standard-height chair, walk 3 meters, turn around, walk back to the chair, and sit down. The total time to complete the task (in seconds) is recorded. Higher times indicate reduced mobility.
  L Test: Time (in seconds) to complete the L-Test of Functional Mobility. The test requires participants to stand up from a chair, walk 3 m, execute a 90° turn, walk another 7 m, perform a 180° turn, and return along the same path (total walking distance ≈ 20 m). The task ends when the participant sits back down. The total time to complete the task (in seconds) is recorded. Higher times indicate reduced mobility.

SUMMARY:
This study aims to investigate the interrater and test-retest reliability of GYKO-based postural sway measurements collected during the L-Test and Timed Up and Go (TUG) test in individuals with Parkinson's disease (Hoehn & Yahr stages 1-3). Two independent raters will perform GYKO-based assessments of the L-Test and TUG with a 20-minute interval. Participants will return one week later to repeat the same procedures for test-retest reliability. Concurrent validity will be examined using the Berg Balance Scale.

DETAILED DESCRIPTION:
This study aims to investigate the test-retest and interrater reliability, as well as the concurrent validity, of GYKO-based postural sway measurements obtained during the L-Test and the Timed Up and Go (TUG) test in individuals with Parkinson's disease. Participants diagnosed with idiopathic Parkinson's disease (Hoehn & Yahr stages 1-3) will be evaluated using the GYKO inertial measurement unit, which provides quantitative postural sway parameters including ellipse area, mean length, mediolateral and anteroposterior mean length, mediolateral and anteroposterior mean distance, and velocity.

Two independent raters will perform GYKO-based assessments of the L-Test and TUG on the same day, with a 20-minute interval between raters, to determine interrater reliability. Participants will return one week later to repeat the same procedures, allowing assessment of test-retest reliability.

To examine concurrent validity, participants' functional balance will also be assessed using the Berg Balance Scale, and correlations between GYKO variables and clinical mobility tests (L-Test and TUG) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Hoehn & Yahr stage 1-3
* Ability to walk independently with or without an assistive device
* Ability to follow verbal instructions
* Age 50-85

Exclusion Criteria:

* Other neurological, vestibular, or musculoskeletal disorders affecting balance
* Deep brain stimulation (DBS) implant
* Severe visual or auditory impairment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 50-85 years with idiopathic Parkinson's disease (Hoehn & Yahr stages 1-3) who can walk independently and participate in TUG, L-Test, and GYKO assessments.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Interrater Reliability of GYKO-Based Postural Sway Parameters | Day 1
  Interrater reliability of postural sway will be evaluated using a composite set of parameters derived from GYKO inertial sensor data collected during the Timed Up and Go (TUG) and L-Test procedures. Measurements will be obtained independently by two raters on the same day.
  The composite postural sway outcome includes ellipsoid area, displacement-related parameters in the mediolateral and anteroposterior directions, and velocity-related parameters. Although individual variables are expressed in different units, all parameters collectively represent a single postural control construct.
  Interrater reliability will be assessed using the intraclass correlation coefficient (ICC 2,1) with 95% confidence intervals.
Test-Retest Reliability of GYKO-Based Postural Sway Parameters | 1 week
  Test-retest reliability of postural sway will be assessed using a composite set of parameters derived from GYKO inertial sensor data collected during the Timed Up and Go (TUG) and L-Test procedures. Participants will be re-evaluated after a 1-week interval.
  The composite postural sway outcome includes ellipsoid area, mediolateral and anteroposterior displacement parameters, and velocity-related parameters, representing a single postural control construct.
  Test-retest reliability will be analyzed using the intraclass correlation coefficient (ICC 3,1) with 95% confidence intervals. Paired t-tests will be used to examine differences between test and retest measurements.

SECONDARY OUTCOMES:
Validity of GYKO Postural Sway Parameters with Functional Mobility (TUG and L-Test) | Day 1
  Concurrent validity will be examined by analyzing the relationship between the composite GYKO-based postural sway parameters obtained during the Timed Up and Go (TUG) and L-Test procedures and functional mobility performance.
  Pearson correlation coefficients will be used to assess the associations between postural sway composite outcomes and TUG and L-Test completion times.
Relationship Between Postural Sway and Balance Performance (Berg Balance Scale) | Day 1
  Balance performance will be assessed using the Berg Balance Scale at baseline. The relationship between Berg Balance Scale scores and the composite GYKO-based postural sway parameters obtained during the Timed Up and Go (TUG) and L-Test procedures will be analyzed using Pearson correlation coefficients.
L test and TUG Completion Time | 1 week
  Functional mobility will be assessed using the Timed Up and Go (TUG) test and the L-Test. The TUG requires participants to stand up from a chair, walk 3 meters, turn, return, and sit down.
  The L-Test is a modified version of the TUG and consists of standing up from a chair, walking 3 meters, performing a 90° turn, walking an additional 7 meters, performing a 180° turn, and returning along the same path (total walking distance approximately 20 meters).
  The time required to complete each test will be recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Akıncı, MSc, Study Chair — Hasan Kalyonuc University; Günseli Usgu, Assoc. Prof., Study Director — Hasan Kalyoncu University; Saadet Nur Çörekçioğlu, P.T., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haas B, Clarke E, Elver L, Gowman E, Mortimer E, Byrd E. The reliability and validity of the L-test in people with Parkinson's disease. Physiotherapy. 2019 Mar;105(1):84-89. doi: 10.1016/j.physio.2017.11.218. Epub 2017 Dec 5. PMID 29395266
- [Background] Zampieri C, Salarian A, Carlson-Kuhta P, Aminian K, Nutt JG, Horak FB. The instrumented timed up and go test: potential outcome measure for disease modifying therapies in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2010 Feb;81(2):171-6. doi: 10.1136/jnnp.2009.173740. Epub 2009 Sep 2. PMID 19726406